CLINICAL TRIAL: NCT02738931
Title: A Phase I, Relative Oral Bioavailability Study of Different Fixed Dose Combinations of Dolutegravir and Lamivudine in Healthy Subjects
Brief Title: Relative Bio-availability Study of Dolutegravir and Lamivudine Fixed Dose Combinations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204993
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: dolutegravir; lamivudine; Bioavailability; fixed dose combinations
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Tablets; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Subject will receive reference treatment DTG 50mg and 3TC 300mg administered as single entity tablets (treatment A) in period 1, experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablet (Product Code AA, treatment B) in period 2 and experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablet (Product Code AB, treatment C) in period 3 in a fasted state. There will be at least 7 days washout between dosing periods.
  Interventions: Drug: Dolutegravir 50 mg tablet; Drug: Lamivudine 300 mg tablet; Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AA); Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AB)
- Treatment Sequence BCA (Experimental): Subject will receive experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablet (Product Code AA, treatment B) in period 1 and experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablet (Product Code AB, treatment C) in period 2 and reference treatment DTG 50mg and 3TC 300mg administered as single entity tablets (treatment A) in period 3 in a fasted state. There will be at least 7 days washout between dosing periods.
  Interventions: Drug: Dolutegravir 50 mg tablet; Drug: Lamivudine 300 mg tablet; Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AA); Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AB)
- Treatment Sequence CAB (Experimental): Subject will receive experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AB, treatment C) in period 1 and reference treatment DTG 50mg and 3TC 300mg administered as single entity tablets (treatment A) in period 2 and experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AA, treatment B) in period 3 in a fasted state. There will be at least 7 days washout between dosing periods.
  Interventions: Drug: Dolutegravir 50 mg tablet; Drug: Lamivudine 300 mg tablet; Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AA); Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AB)
- Treatment Sequence ACB (Experimental): Subject will receive reference treatment DTG 50mg and 3TC 300mg administered as single entity tablets (treatment A) in period 1, experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AB, treatment C) in period 2 and experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AA, treatment B) in period 3 in a fasted state. There will be at least 7 days washout between dosing periods.
  Interventions: Drug: Dolutegravir 50 mg tablet; Drug: Lamivudine 300 mg tablet; Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AA); Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AB)
- Treatment Sequence BAC (Experimental): Subject will receive experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AA, treatment B) in period 1 and reference treatment DTG 50mg and 3TC 300mg administered as single entity tablets (treatment A) in period 2 and experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AB, treatment C) in period 3 in a fasted state. There will be at least 7 days washout between dosing periods.
  Interventions: Drug: Dolutegravir 50 mg tablet; Drug: Lamivudine 300 mg tablet; Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AA); Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AB)
- Treatment Sequence CBA (Experimental): Subject will receive experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AB, treatment C) in period 1 and experimental Dolutegravir/Lamivudine 50 mg/300 mg FDC tablets (Product Code AA, treatment B) in period 2 and reference treatment DTG 50mg and 3TC 300mg administered as single entity tablets (treatment A) in period 3 in a fasted state. There will be at least 7 days washout between dosing periods.
  Interventions: Drug: Dolutegravir 50 mg tablet; Drug: Lamivudine 300 mg tablet; Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AA); Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AB)

INTERVENTIONS:
Drug: Dolutegravir 50 mg tablet — A white, film-coated, round tablet debossed with SV 572 on one side and 50 on the other side. Single dose of one tablet will be administered with 240 mL of water.
Drug: Lamivudine 300 mg tablet — Gray, diamond-shaped tablet, engraved "GX EJ7" on one side and plain on the other side. Single dose of one tablet will be administered with 240 mL of water.
Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AA) — Immediate release oval tablet embossed 'gsk' on one face with white film coat. Single dose of one tablet will be administered with 240 mL of water.
Drug: Dolutegravir/Lamivudine 50 mg/300 mg Tablet (Product Code AB) — Immediate release oval tablet embossed 'gsk' on one face with white film coat. Single dose of one tablet will be administered with 240 mL of water.

SUMMARY:
Dolutegravir (DTG) and lamivudine (3TC) are indicated in combination with other antiretroviral agents for the treatment of human immunodeficiency virus type 1 (HIV-1) infection. Fixed dose combination (FDC) tablets of existing approved drugs are preferred by many patients and offer the potential for increased patient adherence and consequently a reduced likelihood of virological failure and viral resistance.

The purpose of the present study is to evaluate the relative bioavailability of two experimental FDC tablets of DTG and 3TC relative to co-administration of the single entity products in healthy adult subjects.

This study will be conducted as a randomized, open label three-way, crossover design with 6 treatment sequences in approximately 30 subjects. Each subject will have a screening visit within 30 days prior to the first dose of study drug, three treatment periods each with a single dose of study drug and a follow-up visit within 7-14 days after the last dose of study drug. There will be at least 7 days washout between dosing periods. The total duration of participation of a subject in this study will be approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac evaluation (history, electrocardiogram [ECG]).
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilogram (kg) (110 pounds [lbs.)] for men and >= 45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kg/meter square (m^2) (inclusive)
* Male or Female

Female subject of non-reproductive potential: is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

* Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy
* Postmenopausal defined as 12 months of spontaneous amenorrhea; in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

  * Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in protocol.

Exclusion Criteria

* Alanine transaminase (ALT) and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 millisecond (msec)
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and ViiV/GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 1 month prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Creatinine clearance (CrCL) <60 mL/minute (min)
* A positive hepatitis B surface antigen (HBsAg) or a or a positive hepatitis B core antibody with a negative hepatitis B surface antibody, positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
DTG: Area under the concentration-time curve from time 0 extrapolated to infinity (AUC[0-inf]) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for pharmacokinetic (PK) analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
DTG: maximum concentration observed (Cmax) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC: AUC(0-inf) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC: Cmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.

SECONDARY OUTCOMES:
DTG: Area under the concentration-time curve from time 0 to the last measurable timepoint (AUC[0-t]) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
DTG: Drug concentration at 24 hours post-dose (C24) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
DTG: Half-life (t1/2) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
DTG: Absorption lag time (tlag) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
DTG: Time to observed maximal drug concentration (tmax) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
DTG: Apparent oral clearance (CL/F) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of DTG will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC:AUC(0-t) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC: C24 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC:t1/2 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC: tlag | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC: tmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.
3TC: CL/F | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, 24, and 48 hours post-dose
  Serial blood samples for PK analysis of 3TC will be collected. From the plasma concentration-time data, the PK parameters will be determined.
Change from baseline in temperature | Baseline and up to 9 weeks
Change from baseline in systolic and diastolic blood pressure (BP) | Baseline and up to 9 weeks
Change from baseline in pulse rate | Baseline and up to 9 weeks
Number of subjects with adverse events | Up to 9 weeks
Number of subjects with the Toxicity Grade and Change from baseline summary for the Indicated Hematology Parameters | Up to 9 weeks
  The hematology parameters included are platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), neutrophils, lymphocytes, monocytes, eosinophils, basophils.
Number of subjects with the Toxicity Grade and Change from baseline summary for the Indicated Clinical Chemistry Parameters | Up to 9 weeks
  Clinical chemistry parameters included are blood urea nitrogen (BUN), creatinine, glucose, creatine phosphokinase (CPK), potassium, sodium, calcium, AST, ALT, alkaline phosphatase, total and direct bilirubin, total protein, albumin
Number of subjects with urinalysis abnormalities | Up to 9 weeks
  Urinalysis parameters included are specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination (if blood or protein is abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States